CLINICAL TRIAL: NCT05804240
Title: Utility of Three-dimensional Transesophageal Echocardiography in Right Ventricular Function Assessment in Surgical Aortic Valve Replacement, Mini-sternotomy Aortic Valve Replacement, and Transcatheter Aortic Valve Replacement
Brief Title: TEE 3D RV Assessment for SAVR, Mini AVR, and TAVR
Status: Recruiting | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Other Study IDs: iRISID-2022-0802
Record Dates: First submitted 2023-03-07; First posted 2023-04-07 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Right Ventricular Dysfunction
Keywords: Right ventricular dysfunction; Three-dimensional transesophageal echocardiography; Surgical aortic valve replacement; Mini-sternotomy aortic valve replacement; Transcatheter aortic valve replacement
MeSH Terms: conditions — Ventricular Dysfunction, Right

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Surgical aortic valve replacement: Patients who have surgical aortic valve replacement
  Interventions: Diagnostic Test: 3D TEE RVEF
- Mini-sternotomy aortic valve replacement: Patients who have mini-sternotomy aortic valve replacement
  Interventions: Diagnostic Test: 3D TEE RVEF
- Transcatheter aortic valve replacement: Patients who have transcatheter aortic valve replacement
  Interventions: Diagnostic Test: 3D TEE RVEF

INTERVENTIONS:
Diagnostic Test: 3D TEE RVEF — With TEE package software, the investigators measure and calculate 3D TEE RVEF using mid esophageal 4 chamber view

SUMMARY:
Three-dimensional echocardiography has become a gold standard to assess right ventricular (RV) function, and investigators plan to use 3D transesophageal echocardiography to assess RV function in 3 types of aortic valve replacement (AVR): surgical AVR (SAVR), mini-sternotomy AVR (mini AVR), and transcatheter AVR (TAVR).

DETAILED DESCRIPTION:
Objective: Right ventricular (RV) function is known to be a critical factor to determine postoperative outcome in cardiac surgery, and echocardiography plays an important role in RV function assessment. In the previous studies, RV function was reported to be more reduced in surgical aortic valve replacement (SAVR) than transcatheter aortic valve replacement (TAVR), but its assessment was performed by 2-dimensional echocardiography. On the other hand, three-dimensional (3D) echocardiography has been the gold standard to assess RV systolic function (EF: ejection fraction), and its intraoperative use is getting more useful in cardiac surgery given recent technological advance in echocardiography machines. However, realty is that RV function assessment is based on subjective information or traditional RV function indices, mostly due to unfamiliarity of 3D technique.

In this study, the investigators plan to evaluate intraoperative RV function assessment by 3D transesophageal echocardiography (TEE). The investigators will compare 3D RV EF with other traditional RV function indices (RV size, Right Ventricular Index of Myocardial Performance (RIMP), RV fractional area change (FAC), peak systolic velocity of the lateral tricuspid annulus (S'), tricuspid annular plane systolic excursion (TAPSE), speckle tracking echocardiography (STE) in SAVR, mini-sternotomy AVR (mini AVR), and TAVR.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over 18 years old
* Patients who had SAVR, mini AVR, or TAVR

Exclusion criteria:

* Patients' refusal
* Suboptimal echocardiography data for RVEF, RV size, RIMP, RVFAC, TAPSE, S', STE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who had SAVR, mini AVR, and TAVR at Thomas Jefferson University Hospital
Sampling Method: Probability Sample
Enrollment: 78 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
RV function assessment indices with TEE (3D RV EF) | For SAVR and mini AVR, post general anesthesia induction, post cardiopulmonary bypass, and after chest closure, up to the end of procedure. For TAVR, post general anesthesia induction and after valve deployment, up to the end of procedure.
  3D RV EF
RV function assessment indices with TEE (RV size) | For SAVR and mini AVR, post general anesthesia induction, post cardiopulmonary bypass, and after chest closure, up to the end of procedure. For TAVR, post general anesthesia induction and after valve deployment, up to the end of procedure.
  RV size
RV function assessment indices with TEE (RIMP) | For SAVR and mini AVR, post general anesthesia induction, post cardiopulmonary bypass, and after chest closure, up to the end of procedure. For TAVR, post general anesthesia induction and after valve deployment, up to the end of procedure.
  RIMP
RV function assessment indices with TEE (RV FAC) | For SAVR and mini AVR, post general anesthesia induction, post cardiopulmonary bypass, and after chest closure, up to the end of procedure. For TAVR, post general anesthesia induction and after valve deployment, up to the end of procedure.
  RV FAC
RV function assessment indices with TEE (S') | For SAVR and mini AVR, post general anesthesia induction, post cardiopulmonary bypass, and after chest closure, up to the end of procedure. For TAVR, post general anesthesia induction and after valve deployment, up to the end of procedure.
  S'
RV function assessment indices with TEE (TAPSE) | For SAVR and mini AVR, post general anesthesia induction, post cardiopulmonary bypass, and after chest closure, up to the end of procedure. For TAVR, post general anesthesia induction and after valve deployment, up to the end of procedure.
  TAPSE
RV function assessment indices with TEE (STE) | For SAVR and mini AVR, post general anesthesia induction, post cardiopulmonary bypass, and after chest closure, up to the end of procedure. For TAVR, post general anesthesia induction and after valve deployment, up to the end of procedure.
  STE

SECONDARY OUTCOMES:
Postoperative course in days | Postoperative course till patient is discharged from hospital. From date of surgery until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months
  Intubation time (if extubated in OR, it will be 0 day)
ICU stay | From date of surgery until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months
  Postoperative course in days
Hospital stay | From date of surgery until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months
  Postoperative course in days.

CONTACTS AND LOCATIONS:
Overall Officials: Yoshihisa Morita, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lang RM, Badano LP, Mor-Avi V, Afilalo J, Armstrong A, Ernande L, Flachskampf FA, Foster E, Goldstein SA, Kuznetsova T, Lancellotti P, Muraru D, Picard MH, Rietzschel ER, Rudski L, Spencer KT, Tsang W, Voigt JU. Recommendations for cardiac chamber quantification by echocardiography in adults: an update from the American Society of Echocardiography and the European Association of Cardiovascular Imaging. J Am Soc Echocardiogr. 2015 Jan;28(1):1-39.e14. doi: 10.1016/j.echo.2014.10.003. PMID 25559473
- [Result] Ternacle J, Berry M, Cognet T, Kloeckner M, Damy T, Monin JL, Couetil JP, Dubois-Rande JL, Gueret P, Lim P. Prognostic value of right ventricular two-dimensional global strain in patients referred for cardiac surgery. J Am Soc Echocardiogr. 2013 Jul;26(7):721-6. doi: 10.1016/j.echo.2013.03.021. Epub 2013 Apr 25. PMID 23623594
- [Result] Cremer PC, Zhang Y, Alu M, Rodriguez LL, Lindman BR, Zajarias A, Hahn RT, Lerakis S, Malaisrie SC, Douglas PS, Pibarot P, Svensson LG, Leon MB, Jaber WA. The incidence and prognostic implications of worsening right ventricular function after surgical or transcatheter aortic valve replacement: insights from PARTNER IIA. Eur Heart J. 2018 Jul 21;39(28):2659-2667. doi: 10.1093/eurheartj/ehy251. PMID 29741615
- [Result] Kempny A, Diller GP, Kaleschke G, Orwat S, Funke A, Schmidt R, Kerckhoff G, Ghezelbash F, Rukosujew A, Reinecke H, Scheld HH, Baumgartner H. Impact of transcatheter aortic valve implantation or surgical aortic valve replacement on right ventricular function. Heart. 2012 Sep;98(17):1299-304. doi: 10.1136/heartjnl-2011-301203. Epub 2012 Jun 11. PMID 22689711
- [Result] Koo TK, Li MY. A Guideline of Selecting and Reporting Intraclass Correlation Coefficients for Reliability Research. J Chiropr Med. 2016 Jun;15(2):155-63. doi: 10.1016/j.jcm.2016.02.012. Epub 2016 Mar 31. PMID 27330520